CLINICAL TRIAL: NCT05002075
Title: Efficacy of an m-Health Cardiac Rehabilitation Program in Heart Failure With Preserved Ejection Fraction: A Pilot Randomized Controlled Trial
Brief Title: Efficacy of an m-Health Cardiac Rehabilitation Program in Heart Failure With Preserved Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ambarish Pandey, Assistant Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2021-0329
Record Dates: First submitted 2021-07-28; First posted 2021-08-12 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: HFpEF; Cardiac rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care arm (No Intervention): Participants in the usual control group will receive standard of care per their providers' discretion.
- m-health cardiac rehabilitation intervention arm (Experimental): Participants randomized to m-Health cardiac rehabilitation will receive a 24-week home-based exercise program
  Interventions: Other: m-health cardiac rehabilitation

INTERVENTIONS:
Other: m-health cardiac rehabilitation — Participants randomized to m-Health cardiac rehabilitation will receive a 24-week home-based exercise program delivered via a previously validated, commercially available smartphone platform called Movn (Moving Analytics, California). This app includes a patient-facing iOS and Android compatible smartphone app and an integrated hospital-facing online dashboard for remote monitoring and care coordination by a trained coach
  Arms: m-health cardiac rehabilitation intervention arm

SUMMARY:
Heart failure (HF) portends substantial morbidity, mortality, and health care costs in the United States and the prevalence of heart failure with preserved ejection fraction (HFpEF) relative to HF with reduced ejection fraction (HFrEF) has been increasing. HFpEF is associated with a high morbidity and mortality burden and is projected to be the predominant subtype of HF in the near future. While multiple therapies have proven efficacious for patients with HFrEF, no pharmacological agents have demonstrably been shown to improve outcomes in HFpEF, highlighting the need for novel approaches to HFpEF treatment. Exercise intolerance (EI) is the cardinal symptom of HFpEF, which manifests as dyspnea and fatigue. EI leads to functional deconditioning and reduced quality of life (QOL), both of which elevate risk of death and hospitalization in patients with HFpEF. Supervised exercised training is associated with improvements in exercise capacity and QOL in adults with HFpEF. However, supervised exercise has not been widely utilized for the treatment of HFpEF due to logistical and fiscal barriers. Home-based exercise using an m-Health platform is an alternative to supervised exercise that can deliver clinician prescribed exercise interventions and wellness education though monitoring and care coordination. The goal of this study is to evaluate the feasibility and efficacy of a patient specific progressive home-based cardiac rehabilitation program leveraging the technology of the m-Health program in improving functional status, exercise capacity, and QOL in patients with HFpEF.

DETAILED DESCRIPTION:
Approximately 6.2 million adults in the United States suffer from heart failure (HF), of which almost one-half maintain a left ventricle ejection fraction (EF) >50% known as heart failure with preserved ejection fraction (HFpEF). The prevalence of HFpEF has been increasing as compared with HF with reduced ejection fraction (HFrEF) over time, particularly in older adults. HFpEF is associated with a high morbidity and mortality burden and remains recalcitrant to available pharmacotherapies, significantly highlighting the need for novel strategies for management. Emerging data suggests HFpEF is a multiorgan disease with complex pathophysiology culminating in debilitating exercise intolerance (EI). This key clinical manifestation of HFpEF, stems from multiple causal pathways: accelerated fitness decline with aging, high comorbidity burden, sarcopenia, impaired cardiovascular reserve, and skeletal muscle myopathy. EI demonstrated by dyspnea and fatigue cascades into functional deconditioning and reduced quality of life (QOL). In addition to EI, >90% of patients with HFpEF are pre-frail or frail and demonstrate physical function limitations. Unfortunately, these characteristic clinical findings in HFpEF are strongly predictive of death and hospitalization. There is an urgent need to develop effective therapeutic approaches targeting EI and physical function to achieve meaningful improvements in patient-reported and clinical outcomes in HFpEF.

Supervised exercise training has been shown to improve functional status, exercise capacity, quality of life (QOL), and lower risk of hospitalization in patients with HF with most studies conducted in the HFrEF population. Smaller trials have demonstrated significant improvements in exercise capacity and QOL with supervised exercise training in HFpEF.5 Accordingly, the AHA/ACC 2013 HF guidelines recommend exercise and cardiac rehabilitation (CR) for patients with chronic HF who can participate in exercise to improve QOL and functional status. Furthermore, a statement from the AHA committee on exercise, rehabilitation, and prevention recommends exercise intensity, duration, and frequency should be tailored to the individual needs of patients. In 2014, HFrEF became a reimbursable diagnosis for comprehensive cardiac rehabilitation (CR) but HFpEF was excluded due to lack of large-scale clinical end-point driven trial evidence. Despite the established benefits, CR is widely underutilized with <10% of eligible HF participants engaging in the same. CR participation barriers include comprehensive institutional expertise needed, widespread regulations, low reimbursement rates, high patient cost, patient time and travel, and facility requirement. Considering the benefits effects of exercise training on patient-oriented functional outcomes in HFpEF and the lack of availability of the current supervised exercise CR model (3 times/week x 12 weeks) for this patient population, there is a need for a more feasible, scalable, and cost-effective alternative approach to delivering exercise training.

Home-based CR using a m-Health platform is a novel alternative to supervised CR that can deliver clinician specific exercise interventions and CR wellness education with remote monitoring and care coordination. The feasibility and efficacy of home-based CR among patients with HFpEF have not been evaluated but have a critical potential impact for this population. This is particularly relevant given the focus on telehealth and home-based in the era of COVID-19. This represents a significant knowledge gap and opportunity considering the current clinical reality that patients with HFpEF have a high burden of physical function impairment and exercise intolerance, the previously reported benefits of exercise training in this patient population, and the current lack of therapeutic opportunities that can be feasibly implemented on a population scale.

Home-based CR with m-health platform is not the standard of care currently, but is an exploratory intervention.

ELIGIBILITY:
Inclusion criteria:

1. Adults age> 18 years
2. HFpEF with left ventricular ejection fraction >50%
3. Clinically stable and no hospitalization in last 4 weeks
4. Estimated glomerular filtration rate > 45 mL/min/1.73 m2 as measured by the simplified MDRD formula
5. Stable diuretic regimen
6. SPPB <10 or historical (within 12 months) or current Peak (measured or estimated) VO2 <= 60% predicted value for age and gender.

Exclusion criteria:

1. History of cancer or end stage lung disease
2. Estimated glomerular filtration rate < 45 mL/min/1.73 m2 as measured by the simplified MDRD formula
3. Recent HF decompensation
4. Inability to do exercise test
5. Inability to provide written informed consent
6. History of falls

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline Standard physical performance battery score at 3 and 6 months | 3 months and 6 months
  SPPB score is a well-validated measure of physical function using 3 components: 4-m gait speed, time to complete 5 chair rises, and standing balance. Each component is scored on a 0-4 scale and summed for an overall score range of 0-12.

SECONDARY OUTCOMES:
Peak VO2 | 6 months
  Peak VO2 is a gold-standard measure of aerobic exercise capacity and will be measured by maximal exercise test using a previously established ergometer protocol
6-minute walk distance | 3 months and 6 months
  6-MWD is a simple and well-validated measure of submaximal exercise capacity and does not require any exercise equipment or advanced training for technicians
Quality of Life using Kansas City Cardiomyopathy Questionnaire (KCCQ) score | 3 months and 6 months
  QOL will be assessed using the KCCQ score, which is a self-administered questionnaire that assesses a patient's perception of their heart failure with regard to the psychological, physical, and socioeconomic aspects of life. Minimum value is 0 and maximum value is 100. Lower scores means a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Packer M, Fowler MB, Roecker EB, Coats AJ, Katus HA, Krum H, Mohacsi P, Rouleau JL, Tendera M, Staiger C, Holcslaw TL, Amann-Zalan I, DeMets DL; Carvedilol Prospective Randomized Cumulative Survival (COPERNICUS) Study Group. Effect of carvedilol on the morbidity of patients with severe chronic heart failure: results of the carvedilol prospective randomized cumulative survival (COPERNICUS) study. Circulation. 2002 Oct 22;106(17):2194-9. doi: 10.1161/01.cir.0000035653.72855.bf. PMID 12390947
- [Background] Zannad F, McMurray JJ, Krum H, van Veldhuisen DJ, Swedberg K, Shi H, Vincent J, Pocock SJ, Pitt B; EMPHASIS-HF Study Group. Eplerenone in patients with systolic heart failure and mild symptoms. N Engl J Med. 2011 Jan 6;364(1):11-21. doi: 10.1056/NEJMoa1009492. Epub 2010 Nov 14. PMID 21073363
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Background] Lam CSP, Voors AA, de Boer RA, Solomon SD, van Veldhuisen DJ. Heart failure with preserved ejection fraction: from mechanisms to therapies. Eur Heart J. 2018 Aug 7;39(30):2780-2792. doi: 10.1093/eurheartj/ehy301. PMID 29905796
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Background] Pina IL, Apstein CS, Balady GJ, Belardinelli R, Chaitman BR, Duscha BD, Fletcher BJ, Fleg JL, Myers JN, Sullivan MJ; American Heart Association Committee on exercise, rehabilitation, and prevention. Exercise and heart failure: A statement from the American Heart Association Committee on exercise, rehabilitation, and prevention. Circulation. 2003 Mar 4;107(8):1210-25. doi: 10.1161/01.cir.0000055013.92097.40. No abstract available. PMID 12615804
- [Background] Pandey A, MacNamara J, Sarma S, Velasco F, Kannan V, Willard J, Skinner C, Keller T, Basit M, Levine B, Willett D. Rapid-Cycle Implementation of a Multi-Organization Registry for Heart Failure with Preserved Ejection Fraction Using Health Information Exchange Standards. Stud Health Technol Inform. 2019 Aug 21;264:1560-1561. doi: 10.3233/SHTI190534. PMID 31438231
- [Background] Fletcher GF, Ades PA, Kligfield P, Arena R, Balady GJ, Bittner VA, Coke LA, Fleg JL, Forman DE, Gerber TC, Gulati M, Madan K, Rhodes J, Thompson PD, Williams MA; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology, Council on Nutrition, Physical Activity and Metabolism, Council on Cardiovascular and Stroke Nursing, and Council on Epidemiology and Prevention. Exercise standards for testing and training: a scientific statement from the American Heart Association. Circulation. 2013 Aug 20;128(8):873-934. doi: 10.1161/CIR.0b013e31829b5b44. Epub 2013 Jul 22. No abstract available. PMID 23877260
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Popescu BA, Waggoner AD. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2016 Apr;29(4):277-314. doi: 10.1016/j.echo.2016.01.011. No abstract available. PMID 27037982